CLINICAL TRIAL: NCT00403897
Title: An Open Single Centre Study To Assess the Safety and Efficacy of Movicol in the Treatment of Chronic Constipation in Children
Brief Title: An Open Single Centre Study To Assess Treatment of Chronic Constipation in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Dr Mike Geraint, Norgine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99/04
Record Dates: First submitted 2006-11-24; First posted 2006-11-27 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Chronic Constipation
Keywords: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Ages 2 - 6: Day 1= 1 sachet/day; Day 3= 1 sachet BID; Day 5= 1 sachet TID Ages 7 - 11: Day 1= 1 sachet BID; Days 3 & 5 = 2 sachets BID;
  Interventions: Drug: Polyethylene glycol 3350 Na bicarbonate NaCl KCl

INTERVENTIONS:
Drug: Polyethylene glycol 3350 Na bicarbonate NaCl KCl — 6.9g sachet, oral
  Other Names: MOVICOL

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of Movicol in the treatment of chronic constipation in children.

DETAILED DESCRIPTION:
This was a phase III, open, single centre, non-comparative study. All patients were assigned to treatment with Movicol for a period of 12 weeks.

All patients were screened at Day 0 (Visit 1) when baseline assessment of their bowel movements over the previous 14 days were made. Patients were dispensed with Movicol to commence treatment on the following day (Day 1). During the first 5 days the dose was increased on an every second day basis until normal bowel movement was achieved. Thereafter until the end of the study the dosage was titrated according to the stool consistency (diarrhoea, loose stool, hard stools or no bowel movement for 2 days, respectively).

Four on-treatment visits were performed on Day 14 (Visit 2), Day 28 (Visit 3), Day 56 (Visit 4) and Day 84 (Visit 5). At each visit bowel movements over the previous period were assessed by the investigator using the patient's daily diary card data.

ELIGIBILITY:
Inclusion Criteria:

* children aged 24 months - 11 years old inclusive
* patients with constipation defined as:

  * ≤ 2 spontaneous complete bowel movements per week (over the previous 14 days), and one or more of the following:

    * 1/4 or more of bowel movements with straining
    * 1/4 or more of bowel movements with hard or lumpy stools
* patients in whom these symptoms have been present for ≥ 3 months
* new patients or those whose management is unsatisfactory on current laxative treatment
* patients of either sex
* patients of any ethnic origin
* hospital in-patients or outpatients.

Exclusion Criteria:

Patients with:

* history of bowel washout within the last 2 months
* intestinal perforation or history of obstruction
* recent history of urinary tract infection (within last month)
* Hirschsprungs disease
* paralytic ileus
* toxic megacolon
* severe inflammatory conditions of the intestinal tract
* clinically uncontrolled renal/hepatic/cardiac disease(s)
* clinically uncontrolled endocrine disorder(s)
* any other severe unstable co-existing disease
* hypersensitivity to macrogol or other constituents of Movicol
* encopresis
* patients who have taken any investigational drug in the last three months
* patients or patients whose parents would in the opinion of the investigator be unable to comply with the requirements of the study.

Ages: 24 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2001-08; Study Completion 2003-01

PRIMARY OUTCOMES:
The average number of spontaneous complete defaecations per week recorded over the period of treatment between scheduled visits.

SECONDARY OUTCOMES:
Assessment of
abdominal pain
amount of stool
faecal form (Bristol stool scale)
rectal bleeding
pain on defaecation
straining on defaecation
stool withholding
faecal incontinence (soiling)
efficacy (investigator and parental assessment)
concomitant laxative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Winita Hardikar, MD, Principal Investigator — Royal Children's Hospital
Locations (1):
- Royal Children's Hospital, Parkville, Victoria, Australia

REFERENCES:
- [Background] Attar A, Lemann M, Ferguson A, Halphen M, Boutron MC, Flourie B, Alix E, Salmeron M, Guillemot F, Chaussade S, Menard AM, Moreau J, Naudin G, Barthet M. Comparison of a low dose polyethylene glycol electrolyte solution with lactulose for treatment of chronic constipation. Gut. 1999 Feb;44(2):226-30. doi: 10.1136/gut.44.2.226. PMID 9895382